CLINICAL TRIAL: NCT04808414
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Ascending Single and Multiple-Dose Study of the Safety, Tolerability and Pharmacokinetics of Intravenous (IV) QPX9003 in Healthy Adult Subjects
Brief Title: SAD/MAD Safety and PK Study of QPX9003 (Novel Polymyxin) in Normal Healthy Volunteers
Acronym: QPX9003
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qpex Biopharma, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Qpex-300
Record Dates: First submitted 2021-03-16; First posted 2021-03-22 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-07

CONDITIONS: Bacterial Infections
Keywords: polymyxin
MeSH Terms: conditions — Bacterial Infections | interventions — Infusions, Intravenous; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: double-blind, placebo controlled ascending single and multiple dose
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind, placebo controlled ascending single- and multiple-dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- QPX9003 for IV infusion (Experimental): IV novel polymyxin antibiotic Single and Multiple IV doses x 7 days via IV infusion q6hrs
  Interventions: Drug: QPX9003 for IV Infusion
- Placebo for Infusion (Placebo Comparator): IV saline Single and Multiple IV doses x 7 days via IV infusion q6hrs
  Interventions: Drug: Placebo for IV infusion

INTERVENTIONS:
Drug: QPX9003 for IV Infusion — antibiotic
  Other Names: novel IV polymyxin antibiotic
  Arms: QPX9003 for IV infusion
Drug: Placebo for IV infusion — Placebo comparator
  Other Names: IV saline
  Arms: Placebo for Infusion

SUMMARY:
The worldwide spread of resistance to antibiotics among gram-negative bacteria, particularly members of the ESKAPE group of pathogens, has resulted in a crisis in the treatment of hospital acquired infections. In particular, the presence of multi-drug resistant Acinetobacter baumannii and Pseudomonas aeruginosa in hospitals around the world poses a considerable threat.

.

DETAILED DESCRIPTION:
The United States (US) Centers for Disease Control (CDC) have listed multidrug-resistant (MDR) Acinetobacter and MDR Pseudomonas aeruginosa as serious threats [CDC, 2019]. Consistent with the global nature of these resistant bacteria, the World Health Organization (WHO) has designated carbapenem-resistant Acinetobacter baumannii, and carbapenem resistant Pseudomonas aeruginosa as critical threats [WHO, 2017].

To combat these serious threats Qpex has developed QPX9003, a next generation polymyxin that is more potent than existing polymyxins against P. aeruginosa and A. baumannii and has exhibited less nephrotoxicity in preclinical studies.

There remains a significant unmet need for new IV agents to treat gram-negative infections due to resistant bacteria in hospital settings. Some progress has been made in the successful development of new agents to address drug-resistant infections, particularly IV agents for resistant gram-negative bacteria [Talbot et al, 2019]. While some of these agents have addressed urgent threats like carbapenem-resistant Enterobacteriaceae (CRE), their activity is largely confined to strains producing serine carbapenemases; none of these agents have reliable activity against metallo beta-lactamase producing CRE. Moreover, none of these recently approved agents have activity against carbapenem-resistant Acinetobacter baumannii [Talbot et al, 2019]. The increasing prevalence of multidrug-resistant gram-negative bacteria, in particular carbapenemase producing Enterobacteriaceae, A. baumannii, and P. aeruginosa, has resulted in an increase in the use of polymyxin antibiotics as salvage therapy [Biswas et al. 2017].

This Phase 1 study will assess the safety, tolerability and pharmacokinetics of single and multiple IV administered ascending doses (SAD/MAD) of IV QPX9003 in healthy adult subjects.

Qpex is developing IV QPX9003 which is a next generation polymyxin with activity against multi-drug resistant A. baumannii and P. aeruginosa

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males and/or females of non-child bearing potential, 18 to 60 years of age (inclusive).
2. Body mass index (BMI) ≥ 18.5 and ≤ 29.9 (kg/m2) and weight between 55.0 and 100.0 kg (inclusive).
3. Medically healthy with clinically insignificant screening results (e.g., laboratory profiles, medical histories, electrocardiograms [ECGs], physical examination) as assessed by the PI.
4. Voluntarily consent to participate in the study.
5. If male, agree to be sexually abstinent or agree to use a condom when engaging in any sexual activity from Day -1 check-in to the clinic through 30 days following the last administration of the study drug, and to not donate sperm during this same period of time.. If engaging in sexual activity with a female partner of childbearing potential, an additional method of birth control must be used.

   Approved additional methods of birth control include:
   1. Intra-uterine device (IUD) in place for at least 3 months prior to Day 1 through 30 days following the final dosing of the study drug.
   2. Barrier method (diaphragm) for at least 14 days prior to Day 1 through 30 days following the final dosing of the study drug.
   3. Stable hormonal contraceptive for at least 3 months prior to Day 1 through 30 days following the final dosing of the study drug.
   4. Surgical sterilization (vasectomy) at least 6 months prior to Day 1.
6. Females of non-childbearing potential must meet at least one of the following criteria:

   1. postmenopausal (defined as 12 months spontaneous amenorrhea) with a serum FSH leve l≥ 40 mIU/mL.
   2. have undergone one of the following sterilization procedures documented at least 6 months prior to Day 1:

      * Bilateral tubal ligation
      * Hysterectomy
      * Hysterectomy with unilateral or bilateral oophorectomy
      * Bilateral oophorectomy
   3. Females who practice true abstinence or are in same sex relationships where there is no possibility of conception.
7. In addition to meeting Inclusion Criteria 1 through 6, cCohort 12 will consist of normal healthy Chinese subjects who are either:

   a. First generation Chinese subjects born in China, with 2 Chinese biological parents and 4 Chinese grandparents born in China of full Chinese descent.

   i. Subject has lived less than or equal to 10 years outside of China. ii. In addition to mainland China, subjects or their parents and grandparents may also be from Taiwan, Hong Kong, or Mongolia, or b. Second generation Chinese subjects born outside of China with 2 Chinese biological parents and 4 grandparents born in China of full Chinese descent.

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
2. Positive urine drug screen or alcohol breath test at screening or check-in (Day -1).
3. Positive testing for HIV, hepatitis B or C
4. History or presence of alcoholism or drug abuse within last 2 years
5. Use of more than 5 packs/week of tobacco/nicotine-containing product within last 6 months prior dosing.
6. Use of any prescription medication (with the exception of hormonal contraceptives or hormone replacement therapy for females) within 14 days prior to dosing.
7. Use of any over-the-counter (OTC) medication, including herbal products, probiotics and vitamins, within the 7 days prior to dosing.
8. Use of antacids, H2 receptor blockers or proton pump inhibitors 7 days prior to dosing.
9. History of any hypersensitivity reaction or anaphylaxis to any medication, including polymyxin antibiotics.
10. Participation in another investigational clinical trial within 30 days prior to Day 1 or within 5 half-lives of the previous investigational drug, whichever is longer.
11. Females who are pregnant or lactating.
12. QTcF interval >450 msec for males and >470 msec for females, or history of prolonged QT syndrome at screening or check-in.
13. Calculated creatinine clearance less than 80 mL/min (Cockcroft-Gault method) at screening or check-in.
14. Subjects who have any clinically significant abnormalities on laboratory values: White blood cell count < 3,000/mm3, hemoglobin < 11g/dL or Absolute neutrophil count < 1,200/mm3 or platelet count < 120,000/mm3.
15. Liver function abnormalities defined by an elevation in bilirubin, Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) 1.5 x Upper Limit of Normal (ULN) of the normal range for subjects based on age and sex.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment -Emergent Adverse events (AEs) by subject and by cohort (single, multiple and combination dose) | up to 21 days
  Number of patients with Treatment-Emergent AEs by treatment arm, severity and relationship to treatment
Number of patients with changes from baseline in safety parameters (single, multiple and combination dose) | up to 13 days
  Number of patients with changes in safety parameters before and after dosing by subject and treatment arm
Peak plasma Concentration measurements by subject and by cohort (Cmax) (single and combination dose) | up to 13 days
  Comparison will be performed between the cohorts for Cmax. Mean graphical presentation of the data will be reported. Statistical analysis of exposure parameters will be performed.
Area under the plasma concentration versus time curve (AUC) between cohorts (single and multiple dose) | up to 13 days
  Comparison will be performed between the cohorts for AUC. Mean graphical presentation of the data will be reported. Statistical analysis of exposure parameters will be performed.
Urine amount excreted by subject and by cohort (single and combination dose)-PK | up to 13 days
  Urine amount excreted will be calculated from urinary excretion data
Urine % dose excreted by subject and by cohort (single and multiple dose)-PK | up to 13 days
  Urine amount of % dose excreted will be calculated from urinary excretion data

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery S Loutit, MBChB, Study Director — Qpex Biopharma, Inc.
Locations (1):
- Altasciences, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Watkins M, Zhu Y, Griffith DC, Loutit JS, Margolis D, Gu P. Phase 1 study of the safety, tolerability, and pharmacokinetics of a synthetic macrocyclic peptide antibiotic (BRII-693) in healthy adult participants. Antimicrob Agents Chemother. 2025 Jan 31;69(1):e0128824. doi: 10.1128/aac.01288-24. Epub 2024 Dec 9. PMID 39651882